CLINICAL TRIAL: NCT03405051
Title: Hypokalemia in Hospitalized Patients for Heart Failure in the Therapeutic Cardiac Failure Unit: Morbidity-mortality Impact
Brief Title: Hypokalemia in Hospitalized Patients for Heart Failure in the Therapeutic Cardiac Failure Unit
Acronym: HYPIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-03Obs-CHRMT
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure
Keywords: hypokalemia; cardiac failure
MeSH Terms: conditions — Heart Failure; Hypokalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypokalemia is very common in heart failure patients. Deleterious effects have been report on the cardiovascular system. Most of the clinical data concerning this ionic trouble are based on post-hoc study and some findings seemed disjointed.

DETAILED DESCRIPTION:
This study tried to describe hypokalemia impact during hospital stay in hospitalized patients with heart failure and particularly on mortality and re-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in the Therapeutic Cardiac Failure Unit in the CHR Metz-Thionville
* Patient with congestive heart failure

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with congestive heart failure admitted to the Heart Failure Unit in the Mercy hospital (CHR Metz-Thionville).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Composite of death and re-hospitalization | Month 3
  The number of death for any reason and re-hospitalization for congestive heart failure

SECONDARY OUTCOMES:
Death | Month 3
  Percentage of death for any reason
Re-hospitalization | Month 3
  Percentage of re-hospitalization for congestive heart failure
Length of stay | Month 3
  Days spent at the hospital
Incidence of hypokalemia | Month 3
  Percentage of incidence during the stay of hypokalemia
Prevalence of hypokalemia | Month 3
  Percentage of initial prevalence during the stay of hypokalemia

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz-Thionville, Metz, France